CLINICAL TRIAL: NCT02113982
Title: Tagraxofusp in Patients With Acute Myeloid Leukemia (AML) and Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN)
Brief Title: Tagraxofusp in Patients With Blastic Plasmacytoid Dendritic Cell Neoplasm or Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STML-401-0114
Record Dates: First submitted 2014-03-13; First posted 2014-04-15 (Estimated); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN); Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Blastic Plasmacytoid Dendritic Cell Neoplasm; Leukemia, Myeloid, Acute | interventions — tagraxofusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- First-Line Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN) (Experimental): Intervention: Tagraxofusp
  Interventions: Drug: Tagraxofusp
- Relapse/Refractory Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN) (Experimental): Intervention: Tagraxofusp
  Interventions: Drug: Tagraxofusp
- Acute Myeloid Leukemia (Experimental): Intervention: Tagraxofusp
  Interventions: Drug: Tagraxofusp

INTERVENTIONS:
Drug: Tagraxofusp
  Other Names: SL-401

SUMMARY:
This is a 4-stage, non-randomized, open-label, dose escalation and expansion, multicenter study. A cycle of therapy is 21 days. Stage 1 was a dose-escalation stage. During Stages 2-4, patients are treated at the MTD or maximum tested dose at which multiple DLTs are not observed during Stage 1.

DETAILED DESCRIPTION:
Study 0114 is a multi-stage, non-randomized, open-label, multicenter study of Tagraxofusp in First line and Relapsed/Refractory (R/R) Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN) and Acute Myeloid Leukemia (AML) patients divided into 4 stages.

Each study stage has its own unique objectives and patient population, with Stage 1 representing the dose escalation phase and Stage 3 the pivotal phase.

In Stages 1 and 2, both patients with BPDCN (first-line and R/R) and AML were enrolled; Stage 3 enrolled previously untreated (first-line) BPDCN patients only. A separate stage, Stage 4, enrolled First-line and R/R BPDCN patients to further characterize safety and efficacy of Tagraxofusp.

The primary study objectives are reported below by stage:

Stage 1: to determine the Maximum Tolerated Dose (MTD) (or Maximum Tested Dose, MTeD where multiple DLTs were not observed) of Tagraxofusp administered at the following dose levels 7, 9, 12, 16 µg/kg/day

Stage 2: cohort expansion to determine the efficacy and safety of Tagraxofusp at the MTD selected in Stage 1

Stage 3 (pivotal): to determine the efficacy and safety of Tagraxofusp in patients with First-line BPDCN

Stage 4: to further characterize the efficacy and safety of Tagraxofusp in patients with both First-line and R/R BPDCN

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of AML (Protocol Stages 1 and 2) or BPDCN (Protocol Stages 1-4) according to WHO classification (AML; excluding acute promyelocytic leukemia [APL, FAB M3]) or confirmed by hematopathology (BPDCN) (Facchetti et al. 2008).
2. The patient must meet one of the following (a) or (b) or (c):

   1. Has evidence of persistent or recurrent AML (Protocol Stages 1 and 2) in the peripheral blood and/or bone marrow that is refractory to, or has relapsed from, their most recent prior line of treatment.

      * A prior line of treatment is considered an induction regimen if it involves an approved or investigational cytotoxic chemotherapy agent, biological agent, and/or hypomethylating agent administered alone or in a combination regimen, with the intent to induce robust cytoreduction (i.e., CR).
      * The previous induction regimen may have been a SCT with intent to induce a CR.
      * Consolidation and/or maintenance (including SCT) may have been given in CR/CRi, but are not counted as a line of treatment.
      * Hydroxyurea will not be considered a prior line of treatment.
   2. Has previously untreated AML (Protocol Stages 1 and 2) and is considered to be at high risk for disease progression and/or is unlikely to derive more than transient benefit from standard therapy by having at least one of the following:

      * Treatment-related AML, except if it is associated with favorable cytogenetics (e.g., inversion 16, t[16;16], t[8;21], t[15;17]), and not a candidate for SCT in their current disease state.
      * AML with antecedent hematological disease (e.g., MDS, myelofibrosis, polycythemia vera) and not a candidate for SCT.
   3. Has histological and/or cytological evidence of BPDCN by pathologic assessment at the investigative site according to WHO classification (Facchetti et al. 2008) by a pathologist with expertise in hematologic malignancies, that can be measured for treatment response and is either:

      * Previously untreated (i.e., first-line) (Protocol Stages 2-4).
      * Persistent or recurrent in the peripheral blood, bone marrow, spleen, lymph nodes, skin, or other sites after previous treatment with at least 1 line of systemic therapy for BPDCN, e.g., stem cell transplant or chemotherapy (Protocol Stages 1, 2, and 4). A pathology specimen must be available for central pathology review for all BPDCN patients enrolled in Protocol Stages 2-4.
3. The patient is ≥ 18 years old.
4. The patient has an ECOG performance score (PS) of 0-2.
5. The patient has adequate baseline organ function, including cardiac, renal, and hepatic function:

   * Left ventricular ejection fraction (LVEF) ≥ institutional lower limit of normal as measured by MUGA scan or 2-D ECHO within 28 days prior to start of therapy and no clinically significant abnormalities on a 12-lead ECG
   * Serum creatinine ≤ 1.5 mg/dl
   * Serum albumin ≥ 3.2 g/dl
   * Bilirubin ≤ 1.5 mg/dl
   * AST and ALT ≤ 2.5 times the upper limit of normal (ULN)
6. If the patient is a woman of child bearing potential (WOCBP), she has had a negative serum or urine pregnancy test within 1 week prior to treatment.
7. The patient has signed informed consent prior to initiation of any study-specific procedures or treatment.
8. The patient is able to adhere to the study visit schedule and other protocol requirements, including follow-up for survival assessment.
9. The patient (male and female) agrees to use acceptable contraceptive methods for the duration of time on the study, and continue to use acceptable contraceptive methods for 2 months after the last infusion of Tagraxofusp.

Exclusion Criteria:

1. The patient has a diagnosis of acute promyelocytic leukemia (APL; FAB M3).
2. The patient has persistent clinically significant toxicities Grade ≥ 2 from previous chemotherapy (excluding alopecia, nausea, fatigue, and liver function tests (as mandated in the inclusion criteria)).
3. The patient has received treatment with chemotherapy, wide-field radiation, or biologic therapy within 14 days of study entry.
4. The patient has received treatment with another investigational agent within 14 days of study entry.
5. The patient has previously received treatment with Tagraxofusp.
6. The patient has an active malignancy and/or cancer history (excluding AML, BPDCN, or antecedent MDS) that may confound the assessment of the study endpoints. Patients with a past cancer history (within 2 years of entry) with substantial potential for recurrence and/or ongoing active malignancy must be discussed with the Sponsor before study entry. Patients with the following neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ, cervical intraepithelial neoplasia, organ-confined prostate cancer with no evidence of progressive disease.
7. The patient has clinically significant cardiovascular disease (e.g., uncontrolled or any NYHA Class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction or stroke within 6 months of study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication).
8. The patient has uncontrolled, clinically significant pulmonary disease (e.g., COPD, pulmonary hypertension) that in the opinion of the investigator would put the patient at significant risk for pulmonary complications during the study.
9. The patient has known active or suspected CNS leukemia. If suspected, CNS leukemia should be ruled out with relevant imaging and/or examination of cerebrospinal fluid.
10. The patient is receiving immunosuppressive therapy - with the exception of low-dose prednisone (≤ 10 mg/day) - for treatment or prophylaxis of graft-versus-host disease (GVHD). If the patient has been on immunosuppressive treatment or prophylaxis for GVHD, the treatment(s) must have been discontinued at least 14 days prior to study treatment and there must be no evidence of Grade ≥ 2 GVHD.
11. The patient has uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, DIC, or psychiatric illness/social situations that would limit compliance with study requirements.
12. The patient is pregnant or breast feeding.
13. The patient has known positive status for human immunodeficiency virus (HIV) active or chronic Hepatitis B or Hepatitis C.
14. The patient is oxygen-dependent.
15. The patient has any medical condition which in the opinion of the investigator places the patient at an unacceptably high risk for toxicities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2014-09; Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - City of Hope National Medical Center, Duarte, California
  - H. Lee Moffiitt Cancer Center & Research Institute, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center Presbyterian Shady Side, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Konopleva M, Pemmaraju N, Sweet KL, Stein AS, Rizzieri DA, Wang ES, Vasu S, Rosenblat T, Zuurman M, Gupta I, Lane AA. Hematopoietic effects of tagraxofusp in treatment-naive patients with blastic plasmacytoid dendritic cell neoplasm. Cancer. 2026 Jan 1;132(1):e70243. doi: 10.1002/cncr.70243. PMID 41486505
- [Derived] Pemmaraju N, Sweet KL, Stein AS, Wang ES, Rizzieri DA, Vasu S, Rosenblat TL, Brooks CL, Habboubi N, Mughal TI, Kantarjian H, Konopleva M, Lane AA. Long-Term Benefits of Tagraxofusp for Patients With Blastic Plasmacytoid Dendritic Cell Neoplasm. J Clin Oncol. 2022 Sep 10;40(26):3032-3036. doi: 10.1200/JCO.22.00034. Epub 2022 Jul 12. PMID 35820082
- [Derived] Pemmaraju N, Lane AA, Sweet KL, Stein AS, Vasu S, Blum W, Rizzieri DA, Wang ES, Duvic M, Sloan JM, Spence S, Shemesh S, Brooks CL, Balser J, Bergstein I, Lancet JE, Kantarjian HM, Konopleva M. Tagraxofusp in Blastic Plasmacytoid Dendritic-Cell Neoplasm. N Engl J Med. 2019 Apr 25;380(17):1628-1637. doi: 10.1056/NEJMoa1815105. PMID 31018069

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow data and safety data collected by disease, study stage, and dose only. Baseline characteristics data collected by disease and study stage only.
Groups:
- Stage 1 - AML Indication: 7 µg/kg/Day Dosage: All AML study patients who received 7 µg/kg/day of tagraxofusp as IV over 15 minutes for up to 5 consecutive days of a 21-day cycle
- Stage 1 - AML Indication: 9 µg/kg/Day Dosage: All AML study patients who received 9 µg/kg/day of tagraxofusp as IV over 15 minutes for up to 5 consecutive days of a 21-day cycle
- Stage 1 - AML Indication: 12 µg/kg/Day Dosage; Stage 2 - AML Indication: 12 µg/kg/Day Dosage: All AML study patients who received 12 µg/kg/day of tagraxofusp as IV over 15 minutes for up to 5 consecutive days of a 21-day cycle
- Stage 1 - AML Indication: 16 µg/kg/Day Dosage; Stage 2 - AML Indication: 16 µg/kg/Day Dosage: All AML study patients who received 16 µg/kg/day of tagraxofusp as IV over 15 minutes for up to 5 consecutive days of a 21-day cycle
- 1L - Stage 1 - BPDCN Indication: 7 µg/kg/Day Dosage: All BPDCN study patients who received 7 µg/kg/day of tagraxofusp as IV over 15 minutes for up to 5 consecutive days of a 21-day cycle
- 1L - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage; R/R - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage; 1L - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage; R/R - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage; 1L - Stage 3 - BPDCN Indication: 12 µg/kg/Day Dosage; 1L - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage; R/R - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage: All BPDCN study patients who received 12 µg/kg/day of tagraxofusp as IV over 15 minutes for up to 5 consecutive days of a 21-day cycle
Period: Stage 1: Dose Escalation
Arm/Group | Stage 1 - AML Indication: 7 µg/kg/Day Dosage | Stage 1 - AML Indication: 9 µg/kg/Day Dosage | Stage 1 - AML Indication: 12 µg/kg/Day Dosage | Stage 1 - AML Indication: 16 µg/kg/Day Dosage | 1L - Stage 1 - BPDCN Indication: 7 µg/kg/Day Dosage | 1L - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage | Stage 2 - AML Indication: 12 µg/kg/Day Dosage | Stage 2 - AML Indication: 16 µg/kg/Day Dosage | 1L - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage | 1L - Stage 3 - BPDCN Indication: 12 µg/kg/Day Dosage | 1L - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage
Started | 3 | 3 | 2 | 6 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 2 | 6 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 3 | 1 | 0 | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Transplant | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other Therapy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Complicating Disease | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2: Cohort Expansion
Arm/Group | Stage 1 - AML Indication: 7 µg/kg/Day Dosage | Stage 1 - AML Indication: 9 µg/kg/Day Dosage | Stage 1 - AML Indication: 12 µg/kg/Day Dosage | Stage 1 - AML Indication: 16 µg/kg/Day Dosage | 1L - Stage 1 - BPDCN Indication: 7 µg/kg/Day Dosage | 1L - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage | Stage 2 - AML Indication: 12 µg/kg/Day Dosage | Stage 2 - AML Indication: 16 µg/kg/Day Dosage | 1L - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage | 1L - Stage 3 - BPDCN Indication: 12 µg/kg/Day Dosage | 1L - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 34 (Only Stage 2 participants were enrolled into Period 2.) | 1 (Only Stage 2 participants were enrolled into Period 2.) | 13 (Only Stage 2 participants were enrolled into Period 2.) | 10 (Only Stage 2 participants were enrolled into Period 2.) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 1 | 13 | 10 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 0 | 5 | 7 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Transplant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0
Not completed — Patient Preference | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other Therapy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Stage 3: Efficacy Cohort
Arm/Group | Stage 1 - AML Indication: 7 µg/kg/Day Dosage | Stage 1 - AML Indication: 9 µg/kg/Day Dosage | Stage 1 - AML Indication: 12 µg/kg/Day Dosage | Stage 1 - AML Indication: 16 µg/kg/Day Dosage | 1L - Stage 1 - BPDCN Indication: 7 µg/kg/Day Dosage | 1L - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage | Stage 2 - AML Indication: 12 µg/kg/Day Dosage | Stage 2 - AML Indication: 16 µg/kg/Day Dosage | 1L - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage | 1L - Stage 3 - BPDCN Indication: 12 µg/kg/Day Dosage | 1L - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 (Only Stage 3 participants were enrolled into Period 3.) | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Not completed — Transplant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Period: Stage 4: First-line and R/R BPDCN
Arm/Group | Stage 1 - AML Indication: 7 µg/kg/Day Dosage | Stage 1 - AML Indication: 9 µg/kg/Day Dosage | Stage 1 - AML Indication: 12 µg/kg/Day Dosage | Stage 1 - AML Indication: 16 µg/kg/Day Dosage | 1L - Stage 1 - BPDCN Indication: 7 µg/kg/Day Dosage | 1L - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage | Stage 2 - AML Indication: 12 µg/kg/Day Dosage | Stage 2 - AML Indication: 16 µg/kg/Day Dosage | 1L - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage | 1L - Stage 3 - BPDCN Indication: 12 µg/kg/Day Dosage | 1L - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 37 (Only Stage 4 participants were enrolled into Period 4.) | 7 (Only Stage 4 participants were enrolled into Period 4.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 37 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
Not completed — Transplant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Not completed — Radiation Consolidation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Patient Preference | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: modified ITT (mITT): all patients with blastic plasmacytoid dendritic cell neoplasm (first-line or relapsed/refractory) and acute myeloid leukemia who were eligible based on the screening criteria and who received at least 1 dose of tagraxofusp, excluding 2 patients who withdrew from study before first response assessment. Total mITT=136. Baseline characteristics data collected by disease and study stage only.
Groups:
- First-line BPDCN- Stage 1: Dose Escalation, 7 or 12 µg/kg/day of Tagraxofusp as IV over 15 minutes for up to 5 consecutive days of a 21-day cycle
- First-line BPDCN - Stage 2; First-line BPDCN - Stage 3; First-line BPDCN - Stage 4; R/R BPDCN - Stage 2; R/R BPDCN - Stage 4: Administration of 12 µg/kg/day of Tagraxofusp as IV over 15 minutes for up to 5 consecutive days of a 21-day cycle
- R/R BPDCN - Stage 1: Dose Escalation, 12 µg/kg/ day of Tagraxofusp as IV over 15 minutes for up to 5 consecutive days of a 21-day cycle
- AML - Stage 1: Dose Escalation 7, 9,12 or 16 µg/kg/ day of Tagraxofusp as IV over 15 minutes for up to 5 consecutive days of a 21-day cycle
- AML - Stage 2: Administration of 12 µg/kg/ day of Tagraxofusp as IV over 15 minutes for up to 5 consecutive days of a 21-day cycle
- Total: Total of all reporting groups
Arm/Group | First-line BPDCN- Stage 1 | First-line BPDCN - Stage 2 | First-line BPDCN - Stage 3 | First-line BPDCN - Stage 4 | R/R BPDCN - Stage 1 | R/R BPDCN - Stage 2 | R/R BPDCN - Stage 4 | AML - Stage 1 | AML - Stage 2 | Total
Number analyzed (Participants) | 6 | 13 | 13 | 36 | 3 | 10 | 6 | 14 | 35 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10.49) | 62.5 (17.72) | 61.7 (17.15) | 64.1 (14.71) | 72 (7.94) | 69.7 (9.31) | 67.5 (15.32) | 58.6 (11.17) | 61.2 (16.01) | 63.4 (14.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 7 | 0 | 2 | 1 | 7 | 13 | 36
  Male | 5 | 10 | 11 | 29 | 3 | 8 | 5 | 7 | 22 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 12 | 13 | 30 | 2 | 10 | 5 | 12 | 31 | 120
  Other | 1 | 1 | 0 | 6 | 1 | 0 | 1 | 2 | 4 | 16
ECOG Performance Status Scale [Count of Participants; unit: Participants] — Grade 0 Able to carry out all normal activities without restriction.
  Grade 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  Grade 2 Ambulatory and capable of all self-care but unable to carry out any work activities: up and about more than 50% of waking hours.
  Grade 3 Capable of limited self-care; confined to bed or chair more than 50% of waking hours.
  Grade 4 Completely disabled; cannot carry on self-care; totally confined to bed or chair.
  Participants
    ECOG 0 | 3 | 6 | 8 | 16 | 1 | 4 | 2 | 5 | 6 | 51
    ECOG 1 | 3 | 7 | 5 | 17 | 2 | 6 | 4 | 8 | 26 | 78
    ECOG 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 5
    Missing | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: MTD (Stage 1)
Description: Maximum tolerated dose (MTD) in both patients with BPDCN and AML. MTD defined as the highest dose level where less than 2/3 or 2/6 patients experienced a DLT
Time Frame: 21-day period after the first dose (cycle 1)
Population: Patients with First-line Blastic Plasmacytoid Dendritic Cell Neoplasm, R/R Blastic Plasmacytoid Dendritic Cell Neoplasm and Acute Myeloid Leukemia participating to stage 1 (dose-escalation)
Measure: Number; unit: µg/kg/day
Groups:
- First-line BPDCN: First-line BPDCN participants who received at least 1 dose of Tagraxofusp either at 7µg/kg/day or 12 µg/kg/day in stage 1
- R/R BPDCN: R/R BPDCN who received at least 1 dose of Tagraxofusp either at 12 µg/kg/day in Stage 1
- Acute Myeloid Leukemia: AML participants who received at least 1 dose of Tagraxofusp either at 7µg/kg/day, 9 µg/kg/day, 12 µg/kg/day or 16 µg/kg/day in Stage 1
Arm/Group | First-line BPDCN | R/R BPDCN | Acute Myeloid Leukemia
Number analyzed (Participants) | 6 | 3 | 14
µg/kg/day | 12 | 12 | 16

2. Primary Outcome: CR Rate in First-line BPDCN (Stage 3, Pivotal Cohort)
Description: Complete response (CR) rate, defined as the percentage who achieved CR+ CR(clinical) with minimal residual skin abnormality (CRc) after treatment with Tagraxofusp.
  CR criteria according to Cheson BD et al, The International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol 2007;25:579-586:
  Marrow: normalization of blast percentage (≤5%).
  Peripheral blood: normalization of neutrophil count (≥ 1,000/µL) and platelet count (≥ 100,000/µL) - absence of leukemic blasts
  Skin: 100% clearance of all skin lesions from baseline; no new lesions in patients without lesions at baseline
  Nodal masses: regression to normal size on CT
  Spleen, liver: not palpable, nodules disappeared
  CRc criteria: all the above except for skin: marked clearance of all skin lesions from baseline; residual hyperpigmentation or abnormality with BPDCN identified on biopsy (or no biopsy performed)
Time Frame: at pre-defined treatment cycle intervals from randomization up to disease progression, up to 3.5 years
Population: Pre-defined efficacy primary end point assessed in Stage 3, standalone, pivotal efficacy cohort of only patients with first-line BPDCN exposed to 12 μg/kg/day were enrolled.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- First-line BPDCN: First-line blastic plasmacytoid dendritic cell neoplasm (BPDCN) patients enrolled in stage 3
Arm/Group | First-line BPDCN
Number analyzed (Participants) | 13
percentage of participants | 53.8 [25.1 to 80.8]

3. Secondary Outcome: CR Rate in First-line BPDCN, R/R BPDCN and AML
Description: CR rate, defined as the percentage of patients who achieved CR+ CR with minimal residual skin abnormality (CRc) after treatment with Tagraxofusp.
  CR criteria according to Cheson BD et al, The International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol 2007;25:579-586:
  Marrow: normalization of blast percentage (≤5%)
  Peripheral blood: normalization of neutrophil count (≥ 1,000/µL) and platelet count (≥ 100,000/µL) - absence of leukemic blasts
  Skin: 100% clearance of all skin lesions from baseline; no new lesions in patients without lesions at baseline
  Nodal masses: regression to normal size on CT
  Spleen, liver: not palpable, nodules disappeared
  CRc criteria: all the above except for skin: marked clearance of all skin lesions from baseline; residual hyperpigmentation or abnormality with BPDCN identified on biopsy (or no biopsy performed)
Time Frame: at pre-defined treatment cycle intervals from randomization up to disease progression, up to 5 years
Population: Efficacy population including evaluable patients treated at 12 μg/kg/day in the first-line BPDCN, R/R BPDCN and AML.
Measure: Number (95% Confidence Interval); unit: percentage of evaluable patients
Groups:
- First-line BPDCN: First-Line BPDCN patients enrolled across stages
- R/R BPDCN: R/R BPDCN patients enrolled across stages
- Acute Myeloid Leukemia: AML patients enrolled in stage 1-2
Arm/Group | First-line BPDCN | R/R BPDCN | Acute Myeloid Leukemia
Number analyzed (Participants) | 65 | 19 | 36
percentage of evaluable patients | 56.9 [44 to 69.2] | 15.8 [3.4 to 39.6] | 3 [0.1 to 14.2]

4. Secondary Outcome: Duration of CR in First-line BPDCN, R/R BPDCN and AML
Description: Duration of complete response (CR) defined as the time from when the criteria are first met for CR+CRc (whichever was recorded first) until the date that the criteria for relapse after CR+CRc are met, according to the previously reported criteria for CR and CRc and following criteria of relapse after CR+CRc (Cheson BD et al. J Clin Oncol 2007;25:579-586.):
  Marrow: blast percentage >5% (if no peripheral blasts, then confirmation aspirate required ≥ 1week later)
  Peripheral blood: presence of leukemic blasts
  Skin: increase in skin score greater than the sum of nadir plus 50% baseline score
  Nodal masses: appearance of a new lesion(s) >1.5 cm in any axis, ≥50% increase from nadir in SPD of more than one node, or ≥50% increase from nadir in longest diameter of a previously identified node >1cm in short axis
  Spleen, liver: >50% increase from nadir in the SPD of any previous lesions
Time Frame: at pre-defined treatment cycle intervals from randomization up to disease progression, up to 5 years
Population: Efficacy population including evaluable patients treated at 12 μg/kg/day in the first-line BPDCN, R/R BPDCN and AML
Measure: Median (Full Range); unit: months
Groups:
- R/R BPDCN: R/R BPDCN enrolled across stages
- Acute Myeloid Leukemia: AML patients enrolled in stages 1 and 2
Arm/Group | First-Line BPDCN | R/R BPDCN | Acute Myeloid Leukemia
Number analyzed (Participants) | 65 | 19 | 36
months | 24.9 [0.99 to 57.36] | 3.6 [3.02 to 13.93] | 8.6 [NA to NA] — 1 participant only experienced CR

5. Secondary Outcome: ORR in First-line BPDCN, R/R BPDCN and AML
Description: Objective response rate (ORR) defines as the percentage of patients who achieved CR (CR+CRc), CR with incomplete blood count recovery (CRi), or partial response (PR) after treatment with Tagraxofusp according to the previously reported definitions of CR, CRc and the following one of CRi and PR:
  CRi: CR with incomplete of neutrophil and/or platelet count and absence of leukemic blast in the peripheral blood
  Marrow: PR defined as decrease by ≥50% in blast percentage to 5-25%
  Peripheral blood: PR defined as normalization of neutrophil count (≥ 1,000/µL) and platelet count (≥ 100,000/µL)
  Skin: 50%-<100% clearance of all skis lesions from baseline; no new lesions in patients without lesions at baseline
  Nodal masses: ≥50% decrease in SPD of up to 6 largest dominant masses; no increase in size of other nodes
  Spleen, liver: ≥50% in SPD of nodules (for single nodule in greatest transverse diameter); no increase in size of liver or spleen
Time Frame: at pre-defined treatment cycle intervals from randomization up to disease progression, up to 5 years
Population: Efficacy population including evaluable patients treated at 12 μg/kg/day in the first-line BPDCN, R/R BPDCN and AML
Measure: Number (95% Confidence Interval); unit: percentage of evaluable patients
Arm/Group | First-line BPDCN | R/R BPDCN | Acute Myeloid Leukemia
Number analyzed (Participants) | 65 | 19 | 36
percentage of evaluable patients | 75.4 [63.1 to 85.2] | 57.9 [33.5 to 79.7] | 3 [0.1 to 14.2]

6. Secondary Outcome: OS in First-line BPDCN, R/R BPDCN and AML
Description: Overall survival (months) defined as the time from the date of first infusion of Tagraxofusp to the date of death from any cause
Time Frame: From first infusion to treatment discontinuation when survival is assessed every 90 days up to end of follow-up or death, up to 5 years
Population: Efficacy population including evaluable patients treated at 12 μg/kg/day in the first-line BPDCN, R/R BPDCN and AML
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | First-line BPDCN | R/R BPDCN | Acute Myeloid Leukemia
Number analyzed (Participants) | 65 | 19 | 36
Months | 15.8 [9.7 to 25.8] | 8.2 [4.1 to 11.9] | 5.7 [NA to NA] — range 0.49-24 months. 95% CI not estimable

7. Secondary Outcome: Bridge to SCT in First-line BPDCN, R/R BPDCN and AML
Description: Bridge to Stem Cell Transplant (SCT) defined as the percentage of patients who received SCT subsequent to achieving an Investigator-determined outcome from Tagraxofusp that was deemed by the Investigator to enable an SCT
Time Frame: at pre-defined intervals up to achievement of outcome enabling an SCT for a period, up to 5 years
Population: Efficacy population including evaluable patients treated at 12 μg/kg/day in the first-line BPDCN, R/R BPDCN and AML
Measure: Number; unit: percentage of evaluable patients
Arm/Group | First-line BPDCN | R/R BPDCN | Acute Myeloid Leukemia
Number analyzed (Participants) | 65 | 19 | 36
percentage of evaluable patients | 32.3 | 5.3 | 3

ADVERSE EVENTS:
Time Frame: From first dose until 30 days after treatment infusion with the longest treatment exposure of 53.3 months
Description: Considering only 15% of overall patients enrolled across the different stages of the study were treated with dose other than 12µg/kg/day, reporting the adverse events by indication instead of dose level is considered more relevant for safety purpose. The safety population was defined as all patients enrolled in the study who received at least 1 dose of Tagraxofusp; all 138 patients were in the safety population, including 69 first-line BPDCN patients, 20 R/R BPDCN patients, and 49 AML patients.
Arm/Group | Stage 1 - AML Indication: 7 µg/kg/Day Dosage | Stage 1 - AML Indication: 9 µg/kg/Day Dosage | Stage 1 - AML Indication: 12 µg/kg/Day Dosage | Stage 1 - AML Indication: 16 µg/kg/Day Dosage | 1L - Stage 1 - BPDCN Indication: 7 µg/kg/Day Dosage | 1L - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage | Stage 2 - AML Indication: 12 µg/kg/Day Dosage | Stage 2 - AML Indication: 16 µg/kg/Day Dosage | 1L - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage | 1L - Stage 3 - BPDCN Indication: 12 µg/kg/Day Dosage | 1L - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage | R/R - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/2 | 4/6 | 1/3 | 0/3 | 1/3 | 3/34 | 0/1 | 1/13 | 0/10 | 1/13 | 3/37 | 2/7
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 2/2 | 6/6 | 1/3 | 1/3 | 3/3 | 19/34 | 1/1 | 7/13 | 6/10 | 4/13 | 20/37 | 5/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/2 | 6/6 | 3/3 | 3/3 | 3/3 | 34/34 | 1/1 | 13/13 | 10/10 | 13/13 | 37/37 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 - AML Indication: 7 µg/kg/Day Dosage (N=3) | Stage 1 - AML Indication: 9 µg/kg/Day Dosage (N=3) | Stage 1 - AML Indication: 12 µg/kg/Day Dosage (N=2) | Stage 1 - AML Indication: 16 µg/kg/Day Dosage (N=6) | 1L - Stage 1 - BPDCN Indication: 7 µg/kg/Day Dosage (N=3) | 1L - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage (N=3) | R/R - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage (N=3) | Stage 2 - AML Indication: 12 µg/kg/Day Dosage (N=34) | Stage 2 - AML Indication: 16 µg/kg/Day Dosage (N=1) | 1L - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage (N=13) | R/R - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage (N=10) | 1L - Stage 3 - BPDCN Indication: 12 µg/kg/Day Dosage (N=13) | 1L - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage (N=37) | R/R - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 1 | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 4 | 1 | 0 | 1 | 1 | 5 | 2
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Septic Shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Ventricular Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Escherichia Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lactic Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial Paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolic Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival Bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allergic Transfusion Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fluid Overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 - AML Indication: 7 µg/kg/Day Dosage (N=3) | Stage 1 - AML Indication: 9 µg/kg/Day Dosage (N=3) | Stage 1 - AML Indication: 12 µg/kg/Day Dosage (N=2) | Stage 1 - AML Indication: 16 µg/kg/Day Dosage (N=6) | 1L - Stage 1 - BPDCN Indication: 7 µg/kg/Day Dosage (N=3) | 1L - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage (N=3) | R/R - Stage 1 - BPDCN Indication: 12 µg/kg/Day Dosage (N=3) | Stage 2 - AML Indication: 12 µg/kg/Day Dosage (N=34) | Stage 2 - AML Indication: 16 µg/kg/Day Dosage (N=1) | 1L - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage (N=13) | R/R - Stage 2 - BPDCN Indication: 12 µg/kg/Day Dosage (N=10) | 1L - Stage 3 - BPDCN Indication: 12 µg/kg/Day Dosage (N=13) | 1L - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage (N=37) | R/R - Stage 4 - BPDCN Indication: 12 µg/kg/Day Dosage (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 4 | 1 | 1 | 1 | 8 | 0 | 3 | 2 | 3 | 8 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 13 | 0 | 0 | 2 | 3 | 5 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 2 | 1 | 0 | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 3 | 0 | 2 | 1 | 0 | 4 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 4 | 2
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 4 | 0 | 2 | 4 | 1 | 6 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 2 | 2 | 2 | 7 | 0 | 7 | 5 | 5 | 12 | 3
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 6 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 4 | 0 | 0 | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 4 | 0 | 1 | 0 | 3 | 7 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 7 | 0 | 3 | 1 | 5 | 10 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 9 | 0 | 5 | 1 | 2 | 7 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 1 | 0 | 1 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 1 | 2 | 1 | 2 | 1 | 18 | 1 | 8 | 5 | 5 | 13 | 2
Oral mucosa haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 2 | 1 | 0 | 1 | 0
Tongue blistering (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 9 | 1 | 2 | 2 | 3 | 4 | 2
Asthenia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 1 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Chills (General disorders) | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 9 | 0 | 4 | 5 | 2 | 6 | 2
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 2 | 3 | 1 | 0 | 3 | 15 | 1 | 6 | 5 | 7 | 15 | 2
Generalised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 1 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 2 | 1 | 2 | 3 | 0 | 3 | 12 | 0 | 6 | 6 | 4 | 10 | 5
Pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 2 | 2 | 2 | 4 | 1 | 2 | 3 | 12 | 0 | 5 | 6 | 3 | 18 | 1
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 3 | 0 | 2 | 1 | 0 | 1 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 4 | 0 | 0 | 2 | 1 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 2 | 1
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 3 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 3 | 1 | 3 | 2 | 2 | 3 | 20 | 1 | 8 | 5 | 10 | 24 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 2 | 5 | 3 | 2 | 2 | 22 | 1 | 7 | 5 | 9 | 22 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 0 | 3 | 1 | 1 | 1 | 3 | 0 | 0 | 2 | 0 | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 4 | 0 | 2 | 3 | 1 | 3 | 2
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 4 | 0 | 3 | 1 | 1 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 2
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 2 | 0 | 1 | 0 | 1 | 3 | 7 | 1 | 6 | 1 | 6 | 12 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 2 | 0 | 0 | 0 | 2 | 8 | 1 | 3 | 2 | 4 | 4 | 2
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 4 | 1 | 2 | 3 | 7 | 0 | 3 | 3 | 5 | 10 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 4 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 3 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 6 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 0 | 1 | 2 | 0 | 3 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 4 | 3 | 1 | 3 | 21 | 1 | 3 | 8 | 7 | 17 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1 | 3 | 0 | 2 | 2 | 0 | 1 | 2 | 3 | 4 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 8 | 0 | 5 | 2 | 1 | 7 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 2 | 0 | 3 | 4 | 0 | 2 | 1 | 1 | 8 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 4 | 0 | 1 | 2 | 1 | 4 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 5 | 0 | 3 | 3 | 4 | 5 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 3 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 1 | 4 | 1
Dizziness (Nervous system disorders) | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 8 | 0 | 2 | 1 | 3 | 6 | 3
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 11 | 0 | 5 | 1 | 4 | 9 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 0 | 3 | 1 | 2 | 6 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 2 | 3 | 0
Insomnia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 7 | 0 | 3 | 1 | 2 | 3 | 2
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 4 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 5 | 0 | 0 | 2 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 9 | 1 | 1 | 2 | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 10 | 1 | 0 | 3 | 0 | 7 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 9 | 0 | 0 | 1 | 2 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 0 | 1 | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 2 | 0 | 4 | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 5 | 0 | 1 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 2 | 1 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 0 | 4 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 6 | 1 | 1 | 3 | 2 | 8 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Flushing (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 3 | 0 | 2 | 3 | 4 | 3 | 0
Hypotension (Vascular disorders) | 1 | 1 | 2 | 3 | 0 | 0 | 2 | 8 | 1 | 3 | 4 | 4 | 7 | 1

LIMITATIONS AND CAVEATS:
This study was limited by lack of randomization due to the ultra-rare nature of blastic plasmacytoid dendritic cell neoplasm (BPDCN).

Patients lacked established response criteria for BPDCN prior to STML-401-0114.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT02113982/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT02113982/SAP_001.pdf